CLINICAL TRIAL: NCT02044614
Title: Adjuvant Peritoneal Dialysis on a Background of Thrice-Weekly Hemodialysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited patient recruitment
Sponsor: Davita Clinical Research (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DCR-BXT-2013-01
Record Dates: First submitted 2014-01-10; First posted 2014-01-24 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2014-04

CONDITIONS: Functionally Anuric; Hemodialysis/Peritoneal Dialysis
Keywords: Hemodialysis/Peritoneal Dialysis; functionally anuric; Icodextrin; Kidney Disease Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- icodextrin-based peritoneal dialysis to hemodialysis (Other): 12-week course of adjuvant low-frequency icodextrin-based peritoneal dialysis to ongoing thrice-weekly maintenance hemodialysis
  Interventions: Other: Adjuvant Peritoneal Dialysis in the context of ongoing Hemodialysis

INTERVENTIONS:
Other: Adjuvant Peritoneal Dialysis in the context of ongoing Hemodialysis

SUMMARY:
1. To assess the feasibility and safety of applying a 12-week course of adjuvant low-frequency icodextrin-based peritoneal dialysis to an ongoing regimen of thrice-weekly in-center hemodialysis.

   Hypothesis: Icodextrin-based peritoneal dialysis can be safely and feasibly implemented in the context of ongoing thrice-weekly in-center hemodialysis.
2. To measure the effects of a 12-week course of adjuvant low-frequency icodextrin-based peritoneal dialysis to ongoing thrice-weekly maintenance hemodialysis on: inter-hemodialytic weight gain, achievable hemodialytic dry weight, total body water, ambulatory blood pressure, serum phosphorus, and pre-to-post hemodialysis changes in serum potassium and pH, and Kidney Disease Quality of Life-SF physical functioning, energy fatigue, and general health scores.

Hypotheses: Addition of adjuvant icodextrin-based peritoneal dialysis will:

1. reduce inter-hemodialytic weight gain*
2. enable achievement of lower hemodialytic dry weight
3. reduce total body water
4. improve ambulatory blood pressure control
5. reduce serum phosphorus
6. minimize per-hemodialytic changes in serum potassium and pH
7. have favorable effects on indices of physical function and global health

   * Indicates co-primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients who are functionally anuric (urine volume <100ml/day)
* receiving chronic maintenance dialysis for treatment of end-stage renal disease
* transitioning from hemodialysis (HD) to peritoneal dialysis (PD)
* transitioning from PD to HD
* receiving PD and have a functional arteriovenous access already in place

Exclusion Criteria:

* < 18 years of age
* anticipate living related kidney transplant or transfer of care away from a participating unit within the next 6 months
* have anticipated survival <6 months
* have contraindications to PD therapy
* history of complicated bowel or abdominal aortic surgery
* known abdominal wall defects
* pregnancy (including pre-menopausal women not surgically sterilized or on hormonal contraception)
* indwelling trans-abdominal prosthetic devices (e.g., feeding or biliary tubes)
* known hypersensitivity to peritoneal dialysate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Treatment Period (12 weeks)
  Adverse events will be described qualitatively and tabulated by frequency. Levels of icodextrin metabolites (considered individually and in aggregate) will be examined graphically and described in terms of means, standard deviations, medians, inter-quartile ranges, minimums and maximums. In Phase I, the association between Δpre-HD serum osmolality (ie, current pre-HD osmolality-pre-HD osmolality preceding the first icodextrin exchange) and aggregate icodextrin metabolites will be examined graphically and by simple linear regression. The association between pre-to-post-HD changes and serum osmolality and pre-to-post-HD changes in aggregate icodextrin levels will be examined analogously.
baseline-to-follow up changes in inter-HD weight gain | Baseline, before the initiation of icodextrin-based PD, and at the end of the study after 12 weeks of icodextrin-based PD
  Efficacy outcomes will be examined using a self-controlled paradigm considering change in outcome parameters from baseline (ie, on HD alone) to follow up (ie, on HD+PD)
  In most instances, characterization visits will take place following the next hemodialysis treatment, but may be delayed by 1-2 treatments based on pragmatic considerations (appointment availability, day of the week).

SECONDARY OUTCOMES:
baseline-to-follow up changes in HD dry weight (lowest tolerated at each time point) | Baseline, before the initiation of icodextrin-based PD, and at the end of the study after 12 weeks of icodextrin-based PD
  In most instances, characterization visits will take place following the next hemodialysis treatment, but may be delayed by 1-2 treatments based on pragmatic considerations (appointment availability, day of the week).
baseline-to-follow up changes in ambulatory blood pressures | Baseline, before the initiation of icodextrin-based PD, and at the end of the study after 12 weeks of icodextrin-based PD
  In most instances, characterization visits will take place following the next hemodialysis treatment, but may be delayed by 1-2 treatments based on pragmatic considerations (appointment availability, day of the week).
baseline-to-follow up changes in pre-HD serum phosphorus | Baseline, before the initiation of icodextrin-based PD, and at the end of the study after 12 weeks of icodextrin-based PD
  In most instances, characterization visits will take place following the next hemodialysis treatment, but may be delayed by 1-2 treatments based on pragmatic considerations (appointment availability, day of the week).
baseline-to-follow up changes in pre-to-post HD changes in serum potassium and total carbon dioxide (CO2) | Baseline, before the initiation of icodextrin-based PD, and at the end of the study after 12 weeks of icodextrin-based PD
  In most instances, characterization visits will take place following the next hemodialysis treatment, but may be delayed by 1-2 treatments based on pragmatic considerations (appointment availability, day of the week).
baseline-to-follow up changes in Kidney Disease Quality of Life Short Form (KDQoL-SF) scores for physical functioning, energy fatigue, and general health | Baseline, before the initiation of icodextrin-based PD, and at the end of the study after 12 weeks of icodextrin-based PD
  In most instances, characterization visits will take place following the next hemodialysis treatment, but may be delayed by 1-2 treatments based on pragmatic considerations (appointment availability, day of the week).